CLINICAL TRIAL: NCT07243028
Title: Application of Simultaneous Pelvic Floor Ultrasonography and Electromyography Biofeedback on Pelvic Floor Muscle Training
Brief Title: Ultrasound and Electromyography Biofeedback for Pelvic Floor Muscle Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-112-385
Record Dates: First submitted 2025-09-04; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Floor Dysfunction; Pelvic Floor Muscle Weakness
Keywords: Pelvic floor dysfunction; Pelvic floor muscle training; Health behavior; Biofeedback
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Active Comparator): Participants in the ultrasound group received ultrasound-based feedback during the first three sessions, followed by manometry-based feedback during the subsequent three sessions.
  Interventions: Device: Ultrasound Biofeedback Device; Device: Manometer Biofeedback Device
- Manometry Group (Active Comparator): Participants in the manometry group received manometry -based feedback during the first three sessions, followed by ultrasound-based feedback during the subsequent three sessions.
  Interventions: Device: Ultrasound Biofeedback Device; Device: Manometer Biofeedback Device

INTERVENTIONS:
Device: Ultrasound Biofeedback Device — Application of trans-abdominal ultrasonography as a biofeedback tool during pelvic floor muscle training
Device: Manometer Biofeedback Device — Application of manometry as a biofeedback tool during pelvic floor muscle training. The manometer is a routinely used clinical device in hospital-based pelvic floor rehabilitation programs to provide quantitative intravaginal pressure feedback and guide patients in performing correct pelvic floor muscle contractions.

SUMMARY:
This study aims to investigate the factors influencing adherence to pelvic floor muscle training (PFMT) devices among patients with pelvic floor dysfunction (PFD) through structured questionnaires, while simultaneously comparing the effectiveness of different feedback modalities, including non-invasive ultrasound imaging and invasive manometry with electromyography (EMG). By integrating subjective adherence data with objective performance outcomes, the project seeks to evaluate the potential of system-level integration for personalized therapeutic strategies, ultimately enhancing treatment efficacy, improving patient satisfaction, and promoting sustained engagement in PFMT.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 21 years or older diagnosed with pelvic floor muscle dysfunction and requiring pelvic floor muscle training (e.g., for symptomatic pelvic organ prolapse, stress urinary incontinence, or dysfunctional voiding).
2. A Pelvic Floor Disability Index (PFDI-20) score greater than 1.
3. Ability and willingness to provide written informed consent and authorization for the release of personal health information.
4. Willingness and ability to complete all required questionnaires

Exclusion Criteria:

1. Individuals planning a future pregnancy.
2. Inability to read, understand, or sign the written consent form prior to participation.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Bladder base displacement (cm) during pelvic floor muscle contractions measured by transabdominal ultrasound | Baseline and at each of the six pelvic floor muscle training sessions (Sessions 1-6). The six training sessions will be completed within approximately one month, and study parameters will be measured at each of these six sessions by the research staff.
  Transabdominal ultrasound imaging will be employed to provide real-time visualization and quantitative assessment of bladder base displacement during pelvic floor muscle (PFM) contractions. The displacement of the bladder base (in centimeters) will be recorded. Data will be aggregated as mean ± standard deviation.
Change in bladder base angle (degrees) relative to the horizontal line during pelvic floor muscle contractions measured by transabdominal ultrasound | Baseline and at each of the six pelvic floor muscle training sessions (Sessions 1-6). The six training sessions will be completed within approximately one month, and study parameters will be measured at each of these six sessions by the research staff.
  Transabdominal ultrasound imaging will be used to quantify the angular change of the bladder base relative to a horizontal reference line during pelvic floor muscle (PFM) contractions. The angle (in degrees) at rest and during contraction will be recorded, and the difference will be calculated. Data will be summarized as mean ± standard deviation across participants for each session.
Survey on Willingness to Use Pelvic Floor Muscle Training Devices | A total of six pelvic floor muscle training sessions will be completed within approximately one month. Questionnaires will be administered at the 3rd session (midpoint of the treatment) and the 6th session (completion of all training sessions)
  A structured questionnaire designed to assess participants' willingness to use pelvic floor muscle training (PFMT) devices. The survey evaluates multiple domains, including both physical and psychological aspects, providing insights into patient adherence and acceptance of different pelvic floor muscle training (PFMT) assistive tools. The questionnaire is based on a 7-point Likert scale, ranging from 1 ("strongly disagree") to 7 ("strongly agree"). Higher scores indicate greater willingness, acceptance, and positive perception toward the use of pelvic floor muscle training devices.

SECONDARY OUTCOMES:
Surface Electromyography | At each of the six pelvic floor muscle training sessions (Sessions 1-6). The six training sessions will be completed within approximately one month, and outcome parameters will be measured at each of these six sessions by the research staff.
  Electromyographic signals of pelvic floor muscle contractions will be recorded using the wireless surface EMG system.
Vaginal manometry measurement | Measurements will be performed during either the 1st to 3rd sessions (approximately days 1-14 after baseline) or the 4th to 6th sessions (approximately days 15-30 after baseline), according to each participant's assigned randomization sequence.
  A pressure-sensing probe will be inserted vaginally to measure intravaginal pressure (expressed in cmH₂O) generated during pelvic floor muscle contractions.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan